CLINICAL TRIAL: NCT03720301
Title: A Double Blinded, Randomized Controlled Trial of the Use of Osteopathic Medical Manipulation to Decrease the Incidence and Severity of Post-Operative Sore Throat
Brief Title: The Use of Osteopathic Medical Manipulation to Decrease the Incidence and Severity of Post-Operative Sore Throat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kevin Peterson, Anesthesia Resident, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C.2018.129d
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Pharyngitis; Dysphonia
Keywords: Sore Throat; Osteopathic Manipulation; Post operative sore throat; Endotracheal tube
MeSH Terms: conditions — Pharyngitis; Dysphonia | interventions — Manipulation, Osteopathic; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, sham controlled prospective
Who Masked: Participant, Care Provider
Masking Description: Patient and Intubating Anesthesiology provider are blinded to subjects randomization into the sham treatment or protocol treatment arm of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Study arm who will receive pre operative and intraoperative treatments intended to effect POST severity.
  Interventions: Procedure: Osteopathic Manipulation Treatment
- Sham (Sham Comparator): Sham are who will receive a preoperative treatment not intended to effect POST outcomes.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Osteopathic Manipulation Treatment — All techniques with patient supine and physician at head of the bed:
  1. Soft tissue massage to the posterior cervical musculature for approximately 1 minute
  2. Muscle energy to the muscles of neck extension approximately 1 minute
  3. Muscle energy to the Occipital Atlanto (OA) joint 1 minute
  4. Muscle energy to the jaw. Approximately 1 minute
  5. Occipital decompression approximately 1 minute
  6. With time remaining complete another round of soft tissue massage.
  Intraoperative techniques:
  1. Myofascial "Steering wheel" Technique
  2. Sibson's Fascia Release
  3. Occipital decompression
  Arms: Treatment
Procedure: Sham — Sham protocol:
  Patients randomized into the sham arm of the study will undergo a controlled trial tested sham treatment that was shown to induce no statistical improvement in cervical pain or mobility with zero adverse effects with the subjects unable to tell the difference between sham and actual protocol treatment.
  Arms: Sham

SUMMARY:
Post-operative sore throat (POST) ranks as the 8th most undesirable effect in the post-operative period and is noted by up to 90% of patients receiving an endotracheal tube. [1-3] This study aims to show that a simple 5 minute preoperative and intraoperative osteopathic medical manipulation protocol can decrease the severity and or the incidence of post-operative sore throat thereby decreasing morbidity and increasing patient satisfaction and return to daily life.

DETAILED DESCRIPTION:
Subjects are selected in the pre-operative area, based on inclusion criteria the night prior from the operating room list, and given 5 minutes of OMT within 1 hour of intubation and then given a less than 5 minute pre-extubation treatment in the operating room no earlier than 1 hour and no later than 15 minutes prior to expected extubation. The patient will be given a survey to be answered at 1 hour, 6 hours, and 24 hours post operatively. Surveys will be filled out in the hospital by the investigating team electronically or by the subject online after they have departed the hospital (See data collection section for more detail on this procedure). In this manner, the subjects' bias and placebo effect will have limited impact on the study outcomes. There will be randomization tables for men and for women to ensure equal representation of women in both arms of the trial since they bear an independent risk factor by their gender. The intubating anesthesiologist will not know which arm the subject is placed in and will be not be present when the pre-operative treatment is taking place to prevent recognition of sham vs. protocol treatment and possible bias. To accomplish this, treatment will be completed behind a closed curtain. Furthermore, it is unlikely that providers will be able to tell the difference between the sham and protocol treatments if they should see treatment being accomplished. In order to ensure patients meet the 1 hour treatment to intubation criteria patients will be selected from the list of first starts or if they are not on the first start list, treatment will be performed when that patients OR room is in turnover as turnover times average 30+ minutes at this hospital. By performing treatments in this manor there is less risk of OR delays which may prolong treatment to intubation time.

The conduct of the anesthetic is entirely at the discretion of the anesthesia provider but in order to avoid confounding variables there are several requests that will be made concerning the conduct of the anesthetic. If these requests are ignored for the benefit of the patient the subject will be removed from the study as described in this section.

Medications for the induction of anesthesia will be at the provider's discretion, but should include a paralytic and avoid ketamine whenever possible. Use of airway adjuncts such as lidocaine laryngo-tracheal atomizers, lidocaine lollypops, ETT lubrication, etc should be avoided and will result in subject exclusion from this study if used. The exclusion of airway adjuncts is for obvious reasons and the paralytic requirement is to control for subject gag reflex differences that may cause excess trauma to the throat in those with sensitive gag reflexes. Ketamine should be avoided due to the risk of excessive secretions that may result in subject coughing or increased instrumentation with a suction device, and to control for the high analgesia that ketamine might impart to subjects that could skew the data analysis. Use of ketamine during the case will result in removal of the patient from the study, but the lack of paralytic use will not exclude the subject from this study. ETT selection, stylet use, and direct laryngoscopy (DL) blade type/size will be at the provider's discretion. A maximum of 2 intubation attempts will be allowed for subject inclusion into this study to prevent confounding variables of subject anatomy and difficult airways from skewing the data. Only providers with 100 or more intubations should perform intubations on study participants in order to control for poor technique and deviation from this will result in subject removal from the study. ETT cuff pressure should be set at <25cm H2O by aneroid manometer per standard practices. Standard American Society of Anesthesiologists recommended monitors will be employed and maintenance medications will be at provider's discretion with the exception of nitrous oxide which should be avoided due to the potential that it could diffuse into the ETT cuffs causing increased cuff inflation pressure, but will not be a criteria for exclusion from the study. Orogastric and nasogastric tubes should also be avoided as they are a known risk factor for POST but due to the prevalence of their use in this study's potential population their use will not result in study exclusion. Reversal and extubation will be at the provider's discretion with standard extubation criteria and gentle suctioning of oropharyngeal secretions as needed for subject safety. Oropharyngeal suctioning should be avoided if possible due to its link to POST, but its exclusion would pose undue risk of aspiration. Effort should be made to conduct oropharyngeal suctioning as gently as possible. Intraoperative and postoperative analgesics and steroids will be at provider's discretion. All postoperative and intraoperative analgesics will be recorded with time given by the investigative team from the medical record.

No earlier than 1 hour and no later than 15 minutes prior to expected extubation, an additional short OMT session will be conducted in the OR with the subject still anesthetized. The intraoperative session is designed to be less than 5 minutes and will involve minimal to no movement of the subjects head or body so as to not to disturb the surgical team and to prevent the dislodgement of the ETT. Intraoperative treatment is directed at myofascial structures to increase lymphatic and vascular flow to wash away inflammatory products and therefore does not require the subject to be moved or to participate in the treatment. Intra-operative treatment is preferred over post-operative treatment so that inflammatory products can be removed prior to the initial post-operative assessment. Additionally, post-operative treatment sessions could be significantly compromised by patient post-anesthetic agitation/delirium and would require an additional sham treatment to prevent patient un-blinding. There will be no intra-operative treatment for the sham arm of the study to save time and decrease the chance for operative interference. All patients will be told in the recruitment phase that they may receive a second treatment inter-operatively as part of the consent for participation process. Intubation surveys will be conducted prior to the intra-operative treatment session to prevent anesthesia provider bias when they recognize the patient is or is not receiving the second OMT session. At this point there is no further risk of bias to the study by un-blinding the provider.

OMT protocol:

OMT employs many techniques that are either considered direct or indirect techniques. Direct techniques are ones in which the patient is taken into the direction of their motion restriction and then moved further into that motion restriction to move the movement "barrier" toward the normal range of motion end point. Static stretching exercises would be an example of a direct technique. Indirect techniques move the patient away from their motion restriction, or into their "ease" of motion, then aberrant motion barriers are removed by allowing the body to reset myofascial stretch and motion receptors thereby returning them to a balanced range of motion position. An example of an indirect technique would be counterstrain, where in, a muscle that is hypertonic is passively shortened and held until the muscle "relaxes" thereby restoring normal tone. After normal tone is restored the muscle is slowly and passively moved to an anatomically neutral position. Another group of techniques are called myofascial. These are techniques that can be direct or indirect and are focused at the facial layer tissues that surround the lymphatic and vasculature systems with the aim of removing restriction around those vessels so that fluid can flow more freely through them. The protocol used in this study incorporates direct muscle stretching and myofascial techniques that are among some of the most basic and easy to perform.

Protocol treatment:

All techniques with patient supine and physician at head of the bed:

1. Soft tissue massage to the posterior cervical musculature for approximately 1 minute

   * Start with fingers at the cervical thoracic junction and move in rhythmic anterior posterior pattern while pulling cephalad with the fingers in an effort to stretch and relax the paracervical musculature.
2. Muscle energy to the muscles of neck extension approximately 1 minute

   * Passively flex the patient's lower cervical vertebra into the barrier of flexion. With one hand supporting the patients head and one hand palpating the paracervical musculature of the lower cervical spine, have the patient gently extend their neck towards the bed while the physician prevents motion for 3-5 seconds. Then have the patient relax and gently increase the patient's lower cervical flexion once musculature has relaxed completely. Complete 3 rounds of this.
3. Muscle energy to the Occipital Atlanto (OA) joint 1 minute

   * Passively extend the patient's OA joint. With one hand cradling the patients head at the OA joint and the other hand placing two fingers on the patient's forehead. Have the patient flex their head by bringing chin to chest gently with only enough force to flex the muscles of the OA joint. Hold this contraction for 3-5 seconds then gently move the OA further in the extension once the patient relaxes. Complete 3 rounds of this.
4. Muscle energy to the jaw. Approximately 1 minute

   * With patients head resting on a pillow in a sniffing position (lower cervical flexion and OA extension), passively open the patients jaw to the barrier, with one had palpating the muscles of mastication and one to two fingers on the patients chin. Then have the patient gently try to close their mouth against the physician's resistance. Hold for 3-5 seconds than relax. During the relaxation gently move the patients jaw further open. Complete 3 rounds.
5. Occipital decompression approximately 1 minute

   * with patients occiput resting in the palms of the physicians hands gently press the pads of the 2nd through 3rd fingers along the base of the occiput and into the OA joint over the occipital condyles. As the physicians fingers follow along the occiput toward the condyles a gentle outward (lateral) force is applied by bringing the physicians elbow together while continuing to palpate for muscle relaxation. When fingers no longer feel to be "sinking into the neck" (i.e. creep) the treatment is complete.
6. With time remaining complete another round of soft tissue massage.

Intraoperative techniques:

1. Myofascial "Steering wheel" Technique

   * With the physician at the head of the bed the physician places one hand on both of the patient's shoulders over the trapezius muscles with thumbs behind neck and fingers over the clavicles. The physician then palpates down to the facial layer and assess facial motion restrictions in all three planes (anterior/posterior, lateral, rotational). The physician stacks the restrictions either directly or indirectly in all three planes and holds the tissue in this way until there is no more fascial movement or "creep."
2. Sibson's Fascia Release

   * The Physician places the pads of 2nd and 3rd digits over the clavicular notch and applies gentle posterior force to the deep facial layer than applies caudal force directed posterior to the clavicles. As depth increases and creep slows apply a gentle lateral force with each hand and hold until creep is no longer perceived.
3. Occipital decompression

   * Occipital decompression will be performed as described earlier in the preoperative treatment under occipital decompression heading.

Sham protocol:

Patients randomized into the sham arm of the study will undergo a controlled trial tested sham treatment that was shown to induce no statistical improvement in cervical pain or mobility with zero adverse effects with the subjects unable to tell the difference between sham and actual protocol treatment. [16] Below is the same sham treatment protocol used in that study.

1. Movement to the Sham Treatment Position. To move the subject from the neutral position to the sham treatment position, gentle motion is induced by applying pressure to the lateral deltoid region of the subject through the palm of 1 hand while stabilizing the cervical spine with the other hand. This is aimed to induce thoracolumbar side bending with cervical stabilization. To ensure a lack of motion at the cervical spine during the procedure, the cervical-stabilizing hand of the investigator will remain underneath the neck of the subject at all times, isolating the cervical spine from unintended motion during side bending of the thoracolumbar spine by the hand pressing on the lateral deltoid. The hand of the investigator, located beneath the cervical spine while inducing motion, cradles the posterior aspect of the neck, and care will be taken so that the head will not rotate, side bend, or flex.[16]
2. Holding the Subject in the Sham Treatment Position. When the subject is sufficiently side bent such that the opposing shoulder nears the edge of the bed, the hand previously applying force at the lateral deltoid region will be removed, and motion stopped. The hand previously applying force to the lateral deltoid region is then placed at the posterior neck (adjacent to the hand still cupping the posterior neck) to assist in stabilization of the cervical spine, and the subject will rest in this position for 90 seconds.[16]
3. Return to Neutral. The subject will then be returned to midline, again by using gentle lateral shoulder pressure with manual stabilization of the cervical spine; however, in this case, the pressure is applied to the opposite shoulder so that the subject can be returned to the original position. The opposite hand remained beneath the neck of the subject for stabilization, as was done in step 1. [16]

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and over
* ASA class 1, 2, or 3 patients
* BMI <35
* Planned surgery < 2.0 hours

Exclusion Criteria:

* Know difficult airway based on report from patient or review of previous intubation records
* Suspected difficult airway defined as two or more of the following criteria:
* Mallampati 3 or 4
* Mouth opening incisor distance less than 3cm
* Thyromental distance less than 6 cm
* Neck circumference greater than 27 inches
* Surgeries in a position other than supine
* Disease or anatomical abnormalities of the neck, larynx, or pharynx
* Post-operative mechanical ventilation needed
* Nasal intubation
* Active smokers
* Interscalene blocks
* Use of ETT adjuncts (lidocaine LTA, lubrication, etc)
* Ketamine use
* Intubation by provider with less than 100 previous intubations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2018-10-17 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Post Severity | 24 hours
  The primary outcome of this study is a decrease in the severity of Post operative sore throat. Survey questions that are measured at 1, 6, and 24 hours will be analyzed using a 2-way repeated measure ANOVA to compare the 2 randomized arms. All other data including demographic data will be compared using univariate techniques. Categorical data will be summarized using percentages and analyzed using Chi-Squared tests or Fisher's Exact test whichever is most appropriate. Means and standard deviations or medians and inter-quartile ranges will be used as summary statistics for continuous variables and they will be analyzed using Student's t-test or Wilcoxon's Test whichever most appropriate. Significance for results will be established when p-values are less than 0.05.

SECONDARY OUTCOMES:
POST incidence | 24 hours
  Secondary outcome will be a reduction in the cumulative incidence of POST. Analyzed as above.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Peterson, DO, Principal Investigator — Brooke Army Medcial Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No